CLINICAL TRIAL: NCT06640504
Title: Serum Albumin Ratios Correct the Ability of Traditional Biomarkers to Predict Mortality of Sepsis Patients Admitted to Surgical ICU
Brief Title: Serum Albumin Ratios Can Improve Sepsis Mortality Prediction
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Azza Mahrous Shaffik, Lecturer of Anesthesia, Pain & ICU, Benha University
Other Study IDs: Rc 4-9-2024
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients newly admitted to ICU with sepsis or septic shock with manifestations suggestive of sepsis according to the guidelines of the 3rd International consensus definitions for sepsis and septic shock.
  Interventions: Diagnostic Test: serum albumin; Diagnostic Test: C-Reactive Protein; Diagnostic Test: Serum procalcitonin; Drug: Blood Lactate

INTERVENTIONS:
Diagnostic Test: serum albumin — Serum albumin ratios were calculated as the ratio between the estimated blood lactate, and serum levels of CRP and PCT divided by the estimated serum albumin level to get the lactate-to-albumin ratio (LAR), CRP-to-albumin ratio (CAR) and procalcitonin (PCT)-to-albumin ratio (PAR).
Diagnostic Test: C-Reactive Protein — The serum levels of C-reactive protein (CRP) are divided by the estimated serum albumin level to get the CRP-to-albumin ratio (CAR).
Diagnostic Test: Serum procalcitonin — The serum levels of procalcitonin (PCT) are divided by the estimated serum albumin level to get the PCT-to-albumin ratio (PAR).
Drug: Blood Lactate — The serum levels of blood lactate are divided by the estimated serum albumin level to get the lactate-to-albumin ratio (LAR).

SUMMARY:
Sepsis remains a leading cause of mortality in hospitalized patients, despite advancements in critical care. Existing clinical scores for predicting sepsis outcomes often lack generalizability and complexity, hindering accurate risk assessment and timely intervention. This study aimed to evaluate the prognostic performance of serum albumin ratios to C-reactive protein (CRP), procalcitonin (PCT), and lactate in predicting 28-day morbidities and mortality in sepsis patients admitted to surgical ICUs. By incorporating these albumin ratios into clinical decision-making, we hypothesized that clinicians could more accurately identify patients at high risk of adverse outcomes and tailor treatment strategies accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly admitted to ICU with sepsis or septic shock;
* Patients were free of exclusion criteria.

Exclusion Criteria:

* Patients with acute kidney injury;
* Patients with hemorrhagic shock;
* Patients with immunosuppressive or autoimmune disorders;
* Patients suspected to die in ICU.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of all patients admitted to the Surgical Intensive Care Unit with manifestations suggestive of sepsis according to the guidelines of the 3rd International Consensus definitions for sepsis and septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reported having at least a 50% lower risk of mortality in surgical ICU (measured by the APACHE II Scale) in correlation with blood biomarkers ratio. | 1 month
  The diagnostic value of blood biomarkers ratio as lactate-to-albumin ratio (LAR), CRP-to-albumin ratio (CAR), and procalcitonin (PCT)-to-albumin ratio (PAR) in decreased sepsis mortality according to APACHE II Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt